CLINICAL TRIAL: NCT01551680
Title: A Phase I Trial Evaluating Concurrent Whole Brain Radiotherapy and Iniparib (BSI-201) in Multiple Non Operable Brain Metastases
Brief Title: A Trial Evaluating Concurrent Whole Brain Radiotherapy and Iniparib in Multiple Non Operable Brain Metastases
Acronym: RAPIBE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: end of study of this product
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPIBE; 2011-003772-36 (EudraCT Number)
Record Dates: First submitted 2012-02-10; First posted 2012-03-13 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — iniparib

STUDY DESIGN:
Intervention Model Description: Concurrent whole brain radiotherapy and iniparib
Masking Description: Concurrent whole brain radiotherapy and iniparib
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Concurrent whole brain radiotherapy and iniparib (Experimental)
  Interventions: Radiation: Radiation combined with iniparib (BSI-201)

INTERVENTIONS:
Radiation: Radiation combined with iniparib (BSI-201) — Dose escalation of iniparib is implemented according to the CRML method. Three patients will be included at the first dose level (2.8 mg/kg). As long as no DLT is observed, escalation will proceed in cohorts of three patients at least included at the next dose levels (4, 5.6, 8, 11.2 mg/kg). Once a DLT is observed, the CRML will be activated and will be used until the MTD has been found or until six patients have been treated at the highest dose level (11.2 mg/kg). A dose level of 2.0 mg/kg (dose level -1) is included in case the first dose level at 2.8 mg/kg is found to be the MTD.
  Iniparib is given by iv infusion over 1 hour twice weekly. BSI 201 will start the week before the beginning of radiotherapy (W1) and will be continued during the entire irradiation (W2, W3, W4). It will be stopped after 8 injections.
  RT is delivered five days a week over 3 weeks (W2, W3, W4) up to a total dose of 37.5 Gy. Each fraction delivers 2.5 Gy by two opposed tangential fields.

SUMMARY:
Recent pre-clinical and clinical data have indicated that BSI-201 does not possess characteristics typical of the PARP inhibitor class. Based on the results from in vitro and in vivo studies, this trial aims to evaluate the combination of BSI-201 concomitantly with radiotherapy in patients who present with multiple non operable brain metastases. As radiotherapy is a local treatment targeting only the tumor, and because the molecule BSI-201 has shown no major toxicity against tissues without DNA alterations, the proposed combination is expected to provide tumor-selective therapy and leading to a clinical benefit improvement.

Primary objective is to determine the recommended phase II dose (RP2D) and evaluate acute toxicity (CTC-AE v4.0 grading scale) of concurrent administration of whole brain radiotherapy (WBR) and a small molecule BSI-201 in non operable brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Non operable brain metastases from any type of cancer (≥ 2)
* At least one measured brain target available ≥ 1 cm (T1-weighted sequences with contrast application MRI)
* No stereotaxie indication
* Any anterior treatments for systemic disease (any chemotherapy at any line) are accepted but have to be interrupted at least 15 days before and up to 30 days after the present protocol
* No extra-brain disease or stabilized since at least 1 month
* Aged ≥ 18 years old
* KPS > 70 (RPS class I or II)
* Adequate bone marrow function: WBC ≥ 3.5 x 109/L, ANC ≥ 1.5 x 109/L, Platelets ≥ LLN, Hb > 10g/dL,
* Adequate renal function: serum creatinine ≤ 1.5 × ULN and blood urea nitrogen ≤ 25 mg/dL
* Male or female patient using adequate contraceptive method
* Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to the start of treatment
* Informed and signed consent
* Able to be followed according to the terms of the protocol
* Affiliated to the French National social security

Exclusion Criteria:

* Anterior treatment for brain metastases (surgery, radiosurgery, stereotaxie)
* Leptomeningeal metastases
* Inclusion in another protocol within 30 days
* Brain metastases with severe intracranial hypertension clinical signs
* Other cancer except the known primary tumor or in situ cervix cancer or basocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose (MTD) | Until 12 week follow-up
  The MTD is defined as the dose level at which the Dose Limiting Toxicity (DLT) is observed in more than 20% of patients. The DLT is defined as: Any treatment-related toxicity CTC v4.0 ≥ grade 3(CTC-AE v4.0 grading scale)

SECONDARY OUTCOMES:
Rate of adverse events | Until 6 month follow-up
  To evaluate toxicity later than 12 weeks after the end of radiotherapy and iniparib
Quality of life | At baseline, Week 1, Week 4, Week 6, Week 12 and Month 6
  Quality of life will be assessed according to the EORTC QLQ-C30 and QLQ-BN20 questionnaires
Cognitive functions | At baseline, Week 1, Week 4, Week 6, Week 12 and Month 6
  Cognitive functions will be assessed according to the MMS (Mini Mental State) questionnaire
Objective response rate | At 6 and 12 weeks after the end of radiotherapy
  Objective response rates (complete and partial response) will be evaluated by MRI according to the RECIST criteria (v1.1)
Time to local progression | 6 months
  Time to local progression will be measured from the start of treatment until the first date of objectively documented local progression.
Local progression-free survival | 6 months
  Local progression-free-survival will be measured from the start of treatment until the first date of objectively documented local progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: David Azria, MD, PhD, Principal Investigator — CRLC Val d'Aurelle-Paul Lamarque
Locations (3):
- France (3):
  - CRLC Val d'Aurelle-Paul Lamarque, Montpellier
  - AP-HP Hôpital Saint-Louis, Paris
  - Institut Gustave-Roussy, Villejuif